CLINICAL TRIAL: NCT07146399
Title: Ischemic Preconditioning Enhances Autonomic Nervous System Modulation During Frequency Speed of Kick Test in Taekwondo Athletes: A Randomized Crossover Study
Brief Title: The Impact of Ischemic Preconditioning on Exercise Performance and Physiological Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziyue Ou (Other)
Collaborators: Guangzhou Sport University (Other)
Responsible Party: Sponsor-Investigator, Ziyue Ou, Sponsor-Investigator, Guangzhou Sport University
Organization: Guangzhou Sport University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2023LCLL-81
Record Dates: First submitted 2025-08-14; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Preconditioning; Autonomic Nervous System (ANS) Functioning and Mood State
Keywords: Ischemic preconditioning; Autonomic nervous system; Heart rate variability; Heart rate recovery
MeSH Terms: interventions — Ischemic Preconditioning; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPC Trial (Experimental): 220 mmHg
  Interventions: Procedure: Ischemic Preconditioning
- SHAM Trial (Placebo Comparator): 20 mmHg
  Interventions: Procedure: Sham (No Treatment)

INTERVENTIONS:
Procedure: Ischemic Preconditioning — Compression cuff width: 10CM; Compression duration: 5min/5min (ischemia/reperfusion) *4. 220 mmHg
  Arms: IPC Trial
Procedure: Sham (No Treatment) — Compression cuff width: 10CM; Compression duration: 5min/5min (compression/relaxation) *4. 20 mmHg
  Arms: SHAM Trial

SUMMARY:
Ischemic Preconditioning has been confirmed to prevent long-term ischemic damage to tissues, among which the improvement of autonomic nerve system function may be one of its mechanisms of action. In recent years, IPC has gradually been applied to enhance athletic performance and accelerate postexercise recovery; however, there has been limited research on the effects of IPC on ANS function and competitive condition before and after exercise. This study investigated the effects of IPC on ANS function before and after sport-specific testing in taekwondo athletes. The objectives of our study are (1) to investigate the impact of IPC on two indicators of autonomic nervous function-HRV and HRR-and (2) to reveal the coordinating effect of IPC on the sympathetic and parasympathetic nervous systems during the warm-up phase and after specific testing in taekwondo athletes. The investigators hypothesize that IPC enhances sympathetic drive during the warm-up phase and rapidly activates the parasympathetic nervous system postexercise, which is accompanied by improvements in the athletes' competitive condition.

ELIGIBILITY:
Inclusion Criteria:

* Taekwondo athletes with a national ranking of level two or higher, including those placed in the top three at the Provincial Professional Taekwondo Championship (combat) and the top eight at the National Professional Taekwondo Championship (combat);
* adult males aged 18 years or older;
* regular participation in specialized Taekwondo training for the past three months.
* All the subjects were from the same team.

Exclusion Criteria:

* consumption of alcohol or caffeine within 24 hours prior to the experiment;
* engagement in strenuous physical activity within 24 hours before the experiment;
* presence of acute or chronic diseases, including cardiovascular diseases, anxiety disorders, and metabolic diseases;
* use of creatine supplements

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-31 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Taekwondo-specific sports performance test. | Five minutes after the intervention, a standard warm-up lasting 10 minutes is conducted. Following the warm-up, a rest period of 5 minutes is observed. Subsequently, three sets of specialized sports performance tests are administered, with each set lasti
  The specialized athletic ability in Taekwondo is measured by the number of kicks performed during the test.
Heart rate variability | The measurement time points were as follows: heart rate variability was assessed in the resting state upon participants' arrival at the testing site, after a warm-up, and following the sport-specific performance test.
  Used to measure the autonomic nervous function of taekwondo athletes.
Heart rate recovery | The measurement time points were established as follows: heart rate recovery was assessed for 1 minute during the intervals of each test group. Additionally, heart rate recovery was recorded at both 1 minute and 5 minutes following the completion of thre
  Used to measure the autonomic nervous function of taekwondo athletes.
Blood lactate | Blood lactate measurements were taken at several key time points during the study: upon participants' arrival at the test site while they were in a quiet state; at the 3rd minute following the conclusion of the intervention; prior to the commencement of
  Used to measure the intensity and metabolic adaptations during the testing process of taekwondo athletes.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Sport University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The data presented in this study are currently unpublished. The corresponding author will provide the relevant research data upon reasonable request after the associated paper has been officially accepted.

REFERENCES:
- [Background] Tsutsui H, Tanaka R, Yamagata M, Yukimura T, Ohkita M, Matsumura Y. Protective effect of ischemic preconditioning on ischemia/reperfusion-induced acute kidney injury through sympathetic nervous system in rats. Eur J Pharmacol. 2013 Oct 15;718(1-3):206-12. doi: 10.1016/j.ejphar.2013.08.032. Epub 2013 Sep 12. PMID 24036256
- [Background] Lopes TR, Sabino-Carvalho JL, Ferreira THN, Succi JE, Silva AC, Silva BM. Effect of Ischemic Preconditioning on the Recovery of Cardiac Autonomic Control From Repeated Sprint Exercise. Front Physiol. 2018 Oct 26;9:1465. doi: 10.3389/fphys.2018.01465. eCollection 2018. PMID 30416451
- [Background] Noronha Osorio D, Viana-Soares R, Marto JP, Mendonca MD, Silva HP, Quaresma C, Viana-Baptista M, Gamboa H, Vieira HLA. Autonomic nervous system response to remote ischemic conditioning: heart rate variability assessment. BMC Cardiovasc Disord. 2019 Sep 9;19(1):211. doi: 10.1186/s12872-019-1181-5. PMID 31500561
- [Background] Murry CE, Jennings RB, Reimer KA. Preconditioning with ischemia: a delay of lethal cell injury in ischemic myocardium. Circulation. 1986 Nov;74(5):1124-36. doi: 10.1161/01.cir.74.5.1124. PMID 3769170